CLINICAL TRIAL: NCT02687412
Title: Fast-track Surgery After Gynaecological Oncological Surgery
Brief Title: Fast-track Surgery After Gynecological Oncology Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ling Cui (Other)
Responsible Party: Sponsor-Investigator, Ling Cui, MD, Sichuan Cancer Hospital and Research Institute
Organization: Sichuan Cancer Hospital and Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SichuanCHRI
Record Dates: First submitted 2016-02-02; First posted 2016-02-22 (Estimated); Results first posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-08

CONDITIONS: Length of Stay; Postoperative Complications; CRP
Keywords: Fast-track surgery; Gynecological oncology; Hospitalization post-operation; Complication
MeSH Terms: conditions — Postoperative Complications | interventions — Counseling; Educational Status; Cathartics; Carbohydrates

STUDY DESIGN:
Intervention Model Description: prospective randomised controlled trial
Masking Description: Patients were randomly divided into two groups（ FTS group/traditional group）, after that doctors and patients were aware of the grouping situation.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fast-track Surgery (Experimental): Pre-operative: Assessment, counseling and education; preoperative nutritional drink up to 4 h prior to surgery, bowel preparation, only oral intestinal cleaner，antimicrobial prophylaxis and skin preparation; preoperative treatment with carbohydrates (patients without diabetes). Intraoperative : fast solid food before 6 h and liquid food Intake of clear fluids 2 h before anaesthesia; avoiding hypothermia keeping temperature at 36 ±0.5℃, antiemetics at end of anaesthesia. Post-operative : Postoperative glycaemic control; postoperative nausea and vomiting (PONV) control; early postoperative diet(3-6 h after surgery).
  Interventions: Procedure: pre-operative assessment, counseling and education; Procedure: Preoperative nutritional drink up to 4 h prior to surgery; Procedure: bowel preparation; Procedure: preoperative treatment with carbohydrates; Procedure: fast solid; Procedure: avoiding hypothermia; Procedure: Postoperative glycaemic control; Procedure: postoperative nausea and vomiting (PONV) control;; Procedure: early postoperative diet
- Traditional surgery (Other): pre-operative assessment：pre-operative fasting at least 8h, bowel preparation for traditional surgery, Antimicrobial prophylaxis and skin preparation or mechanical bowl until liquid stool Intraoperative: keeping the intra-operative lowtemperature at 34.7±0.6 degree centigrade.
  Post-operative: 6 h after surgery, patients resumed a liquid diet, patients began to take solid diet after anal exhaust
  Interventions: Procedure: pre-operative fasting at least 8h; Procedure: bowel preparation for traditional surgery; Procedure: began to take solid diet after anal exhaust

INTERVENTIONS:
Procedure: pre-operative assessment, counseling and education — pre-operative assessment, counseling and FT management education
  Arms: Fast-track Surgery
Procedure: Preoperative nutritional drink up to 4 h prior to surgery — Preoperative nutritional drink up to 4 h prior to surgery mechanical bowl preparation should not be used
  Arms: Fast-track Surgery
Procedure: bowel preparation — patients are not received mechanical bowel preparation, only oral intestinal cleaner 12 h pre-operation can be accepted, but no need of liquid stool
  Arms: Fast-track Surgery
Procedure: preoperative treatment with carbohydrates — preoperative treatment with carbohydrates (patients without diabetes).
  Arms: Fast-track Surgery
Procedure: fast solid — fast solid food before 6 h and liquid food Intake of clear fluids 2 h before anaesthesia;
  Arms: Fast-track Surgery
Procedure: avoiding hypothermia — avoiding hypothermia, keeping the intra-operative lowtemperature at 36 ±0.5 degree centigrade; antiemetics at end of anaesthesia.
  Arms: Fast-track Surgery
Procedure: Postoperative glycaemic control — Postoperative glycaemic control;
  Arms: Fast-track Surgery
Procedure: postoperative nausea and vomiting (PONV) control;
  Arms: Fast-track Surgery
Procedure: early postoperative diet — early postoperative diet(3-6 h after surgery, patients resumed a liquid diet, 12 h after surgery patients began to take solid diet).
  Arms: Fast-track Surgery
Procedure: pre-operative fasting at least 8h
  Arms: Traditional surgery
Procedure: bowel preparation for traditional surgery — Oral bowel preparations or mechanical bowl until liquid stool
  Arms: Traditional surgery
Procedure: began to take solid diet after anal exhaust — 6 h after surgery, patients resumed a liquid diet, patients began to take solid diet after anal exhaust
  Arms: Traditional surgery

SUMMARY:
Fast-track surgery (FTS) pathway, also known as enhanced recovery after surgery (ERAS), FTS is a multidisciplinary approach aiming to accelerate recovery, reduce complications, minimize hospital stay without an increased readmission rate and reduce healthcare costs, all without compromising patient safety. It has been used successfully in non-malignant gynecological surgery, but it has been proven to be especially effective in elective colorectal surgery. However, no consensus guideline has been developed for gynecological oncology surgery although surgeons have attempted to introduce slightly modified FTS programmes for patients undergoing such surgery. NO randomised controlled trials for now.

The advantages of fast-track most likely extend to gynecology, although so far have scarcely been reported. There is a existing research showed FTS in gynecological oncology provide early hospital discharge after gynaecological surgery meanwhile with high levels of patient satisfaction.

The aim of this study is to identify patients following a FTS program who have been discharged earlier than anticipated after major gynaecological/gynaecological oncologic surgery and analyze the complication after surgery.

DETAILED DESCRIPTION:
Methods/Design

Comparison of Fast-Track (FT) and traditional management protocols. the primary endpoints is length of hospitalization post-operation (d, mean±SD). It was calculated by the difference between date of discharge and date of surgery. The secondary endpoints are complications in both groups are assessed during the first 21 days postoperatively. Including infection(wound infection, lung infection, intraperitoneal infection, operation space infection), postoperative nausea and vomiting (PONV) , ileus, postoperative hemorrhage, postoperative thrombosis and APACHE II score.

The advantages of fast-track most likely extend to gynecology, although so far have scarcely been reported. NO randomised controlled trials for now. The aim of this study is to compare the LOS (Length of hospitalization post-operation) after the major gynaecological/gynaecological oncologic surgery and analyze the complication after surgery. This trial can show whether the FTS program can achieve early hospital discharge after gynaecological surgery meanwhile with low levels of complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for gynecological oncology surgery(including radical hysterectomy add lymphadenectomy, hysterectomy add lymphadenectomy and cytoreductive)
2. Aged 18 years or older
3. Signed informed consent provided

Exclusion Criteria:

1. Patients with a documented infection at the time of operation
2. Aged 71 years or older
3. Patients with ileus at the time of operation
4. Patients with hypocoagulability
5. Patients with psychosis, Alcohol dependence or drug abuse history
6. Patients with primary nephrotic or hepatic disease
7. Patients with severe hypertension systolic pressure≥160mmHg, diastolic pressure>90mmHg

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2017-09-02 (Actual); Study Completion 2018-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ling Cui, MD, Study Chair — Sichuan Cancer Hospital and Research Institute; Yu Shi, Principal Investigator — Sichuan Cancer Hospital and Research Institute; Hong Liu, Principal Investigator — Sichuan Cancer Hospital and Research Institute; Dengfeng Wang, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (1):
- LinShuangfeng, Leshan, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kehlet H. Fast-track colorectal surgery. Lancet. 2008 Mar 8;371(9615):791-3. doi: 10.1016/S0140-6736(08)60357-8. No abstract available. PMID 18328911
- [Background] Kehlet H, Wilmore DW. Multimodal strategies to improve surgical outcome. Am J Surg. 2002 Jun;183(6):630-41. doi: 10.1016/s0002-9610(02)00866-8. PMID 12095591
- [Background] Polle SW, Wind J, Fuhring JW, Hofland J, Gouma DJ, Bemelman WA. Implementation of a fast-track perioperative care program: what are the difficulties? Dig Surg. 2007;24(6):441-9. doi: 10.1159/000108327. Epub 2007 Sep 13. PMID 17851238
- [Result] Acheson N, Crawford R. The impact of mode of anaesthesia on postoperative recovery from fast-track abdominal hysterectomy: a randomised clinical trial. BJOG. 2011 Feb;118(3):271-3. doi: 10.1111/j.1471-0528.2010.02811.x. No abstract available. PMID 21226823
- [Result] Bardram L, Funch-Jensen P, Jensen P, Crawford ME, Kehlet H. Recovery after laparoscopic colonic surgery with epidural analgesia, and early oral nutrition and mobilisation. Lancet. 1995 Mar 25;345(8952):763-4. doi: 10.1016/s0140-6736(95)90643-6. PMID 7891489
- [Result] Carter J, Szabo R, Sim WW, Pather S, Philp S, Nattress K, Cotterell S, Patel P, Dalrymple C. Fast track surgery: a clinical audit. Aust N Z J Obstet Gynaecol. 2010 Apr;50(2):159-63. doi: 10.1111/j.1479-828X.2009.01134.x. PMID 20522073
- [Result] Bona S, Molteni M, Rosati R, Elmore U, Bagnoli P, Monzani R, Caravaca M, Montorsi M. Introducing an enhanced recovery after surgery program in colorectal surgery: a single center experience. World J Gastroenterol. 2014 Dec 14;20(46):17578-87. doi: 10.3748/wjg.v20.i46.17578. PMID 25516673
- [Result] Carter J. Fast-track surgery in gynaecology and gynaecologic oncology: a review of a rolling clinical audit. ISRN Surg. 2012;2012:368014. doi: 10.5402/2012/368014. Epub 2012 Dec 24. PMID 23320193
- [Result] Fearon KC, Ljungqvist O, Von Meyenfeldt M, Revhaug A, Dejong CH, Lassen K, Nygren J, Hausel J, Soop M, Andersen J, Kehlet H. Enhanced recovery after surgery: a consensus review of clinical care for patients undergoing colonic resection. Clin Nutr. 2005 Jun;24(3):466-77. doi: 10.1016/j.clnu.2005.02.002. Epub 2005 Apr 21. PMID 15896435
- [Result] Kehlet H. Multimodal approach to postoperative recovery. Curr Opin Crit Care. 2009 Aug;15(4):355-8. doi: 10.1097/MCC.0b013e32832fbbe7. PMID 19617822
- [Result] Kehlet H. Fast-track surgery-an update on physiological care principles to enhance recovery. Langenbecks Arch Surg. 2011 Jun;396(5):585-90. doi: 10.1007/s00423-011-0790-y. Epub 2011 Apr 6. PMID 21468643
- [Result] Kehlet H, Wilmore DW. Evidence-based surgical care and the evolution of fast-track surgery. Ann Surg. 2008 Aug;248(2):189-98. doi: 10.1097/SLA.0b013e31817f2c1a. PMID 18650627
- [Result] Kranke P, Redel A, Schuster F, Muellenbach R, Eberhart LH. Pharmacological interventions and concepts of fast-track perioperative medical care for enhanced recovery programs. Expert Opin Pharmacother. 2008 Jun;9(9):1541-64. doi: 10.1517/14656566.9.9.1541. PMID 18518784
- [Result] Lin YS. Preliminary results of laparoscopic modified radical hysterectomy in early invasive cervical cancer. J Am Assoc Gynecol Laparosc. 2003 Feb;10(1):80-4. doi: 10.1016/s1074-3804(05)60239-3. PMID 12554999
- [Result] Lu D, Wang X, Shi G. Perioperative enhanced recovery programmes for gynaecological cancer patients. Cochrane Database Syst Rev. 2015 Mar 19;2015(3):CD008239. doi: 10.1002/14651858.CD008239.pub4. PMID 25789452
- [Result] Lv D, Wang X, Shi G. Perioperative enhanced recovery programmes for gynaecological cancer patients. Cochrane Database Syst Rev. 2010 Jun 16;(6):CD008239. doi: 10.1002/14651858.CD008239.pub2. PMID 20556792
- [Result] Marx C, Rasmussen T, Jakobsen DH, Ottosen C, Lundvall L, Ottesen B, Callesen T, Kehlet H. The effect of accelerated rehabilitation on recovery after surgery for ovarian malignancy. Acta Obstet Gynecol Scand. 2006;85(4):488-92. doi: 10.1080/00016340500408325. PMID 16612713
- [Result] Moher D, Schulz KF, Altman DG; CONSORT GROUP (Consolidated Standards of Reporting Trials). The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomized trials. Ann Intern Med. 2001 Apr 17;134(8):657-62. doi: 10.7326/0003-4819-134-8-200104170-00011. PMID 11304106
- [Result] Mortensen K, Nilsson M, Slim K, Schafer M, Mariette C, Braga M, Carli F, Demartines N, Griffin SM, Lassen K; Enhanced Recovery After Surgery (ERAS(R)) Group. Consensus guidelines for enhanced recovery after gastrectomy: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Br J Surg. 2014 Sep;101(10):1209-29. doi: 10.1002/bjs.9582. Epub 2014 Jul 21. PMID 25047143
- [Result] Philp S, Carter J, Pather S, Barnett C, D'Abrew N, White K. Patients' satisfaction with fast-track surgery in gynaecological oncology. Eur J Cancer Care (Engl). 2015 Jul;24(4):567-73. doi: 10.1111/ecc.12254. Epub 2014 Oct 21. PMID 25335828
- [Result] Pruthi RS, Nielsen M, Smith A, Nix J, Schultz H, Wallen EM. Fast track program in patients undergoing radical cystectomy: results in 362 consecutive patients. J Am Coll Surg. 2010 Jan;210(1):93-9. doi: 10.1016/j.jamcollsurg.2009.09.026. Epub 2009 Oct 28. PMID 20123338
- [Result] Sjetne IS, Krogstad U, Odegard S, Engh ME. Improving quality by introducing enhanced recovery after surgery in a gynaecological department: consequences for ward nursing practice. Qual Saf Health Care. 2009 Jun;18(3):236-40. doi: 10.1136/qshc.2007.023382. PMID 19468009
- [Derived] Chau JPC, Liu X, Lo SHS, Chien WT, Hui SK, Choi KC, Zhao J. Perioperative enhanced recovery programmes for women with gynaecological cancers. Cochrane Database Syst Rev. 2022 Mar 15;3(3):CD008239. doi: 10.1002/14651858.CD008239.pub5. PMID 35289396
- [Derived] Cui L, Shi Y, Zhang GN. Fast-track surgery after gynaecological oncological surgery: study protocol for a prospective randomised controlled trial. Trials. 2016 Dec 15;17(1):597. doi: 10.1186/s13063-016-1688-3. PMID 27978842

RESULTS

PARTICIPANT FLOW:
Groups:
- Fast-track Surgery: Pre-operative: pre-operative assessment, counseling and FT management education; preoperative nutritional drink up to 4 h prior to surgery; mechanical bowl preparation should not be used; patients are not received mechanical bowel preparation, only oral intestinal cleaner 12 h pre-operation can be accepted, but no need of liquid stool; antimicrobial prophylaxis and skin preparation; preoperative treatment with carbohydrates (patients without diabetes).
  Intraoperative : fast solid food before 6 h and liquid food Intake of clear fluids 2 h before anaesthesia; avoiding hypothermia, keeping the intra-operative lowtemperature at 36 ±0.5 degree centigrade; antiemetics at end of anaesthesia.
  Post-operative : Postoperative glycaemic control; postoperative nausea and vomiting (PONV) control; early postoperative diet(3-6 h after surgery, patients resumed a liquid diet, 12 h after surgery patients began to take solid diet).
- Traditional Surgery: pre-operative assessment：pre-operative fasting at least 8h, oral bowel preparation or, Antimicrobial prophylaxis and skin preparation or mechanical bowl until liquid stool Intraoperative: keeping the intra-operative lowtemperature at 34.7±0.6 degree centigrade.
  Post-operative: 6 h after surgery, patients resumed a liquid diet, patients began to take solid diet after anal exhaust
  pre-operative fasting at least 8h
  Oral bowel preparations: Oral bowel preparations or mechanical bowl until liquid stool
  intra-operative lowtemperature at 34.7 ±0.6 degree centigrade: keeping the intra-operative lowtemperature at 34.7 ±0.6 degree centigrade
  began to take solid diet after anal exhaust: 6 h after surgery, patients resumed a liquid diet, patients began to take solid diet after anal exhaust
Period: Overall Study
Arm/Group | Fast-track Surgery | Traditional Surgery
Started | 50 | 57
Completed | 50 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients scheduled for gynaecological oncology surgery (including radical hysterectomy and lymphadenectomy, hysterectomy and lymphadenectomy, and cytoreductive procedures for both open and laparoscopic surgery)
Groups:
- Total: Total of all reporting groups
Arm/Group | Fast-track Surgery | Traditional Surgery | Total
Number analyzed (Participants) | 50 | 57 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 53 | 100
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (9.70) | 50 (10.52) | 49 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 57 | 107
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 50 | 57 | 107
Body surface area [Mean (Standard Deviation); unit: m^2] | 1.5462 (0.11873) | 1.5362 (0.11550) | 1.5409 (0.11658)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 22.681 (4.1774) | 23.165 (3.2728) | 22.939 (3.7722)

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospitalization Post-operation
Description: days from operation date to discharge date
Time Frame: up to 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fast-track Surgery | Traditional Surgery
Number analyzed (Participants) | 50 | 57
days | 8.92 (2.029) | 9.67 (3.119)
Statistical Analysis 1: Comparison: Fast-track Surgery vs Traditional Surgery; Test type: Superiority; p = 0.141, t-test, 2 sided

2. Primary Outcome: The Total Cost (RMB)
Description: The total cost from hospitalization
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: RMB
Arm/Group | Fast-track Surgery | Traditional Surgery
Number analyzed (Participants) | 50 | 57
RMB | 38882.44 (8557.800) | 42864.12 (10166.535)
Statistical Analysis 1: Comparison: Fast-track Surgery vs Traditional Surgery; Test type: Superiority; p = 0.029, t-test, 2 sided; Mean Difference (Final Values) = -4041, 95% CI 2-sided [-7672.301 to -411.065], Standard Error of Mean 1831.042

3. Secondary Outcome: CRP
Description: C-Reactive protein mg/L
Time Frame: up to 12 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Fast-track Surgery | Traditional Surgery
Number analyzed (Participants) | 50 | 57
mg/L | 42.125 (28.4284) | 62.499 (37.7870)
Statistical Analysis 1: Comparison: Fast-track Surgery vs Traditional Surgery; Test type: Superiority; p = 0.002, t-test, 2 sided; Mean Difference (Final Values) = 20.3739, 95% CI 2-sided [7.6414 to 33.1065], Standard Error of Mean 6.4198

4. Secondary Outcome: Number of Participants With Complications
Description: Count of patients with complications in both groups are assessed during the first 21 days postoperatively. Including infection(wound infection, lung infection, intraperitoneal infection, operation space infection), postoperative nausea and vomiting (PONV) , ileus, postoperative hemorrhage, postoperative thrombosis.
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fast-track Surgery | Traditional Surgery
Number analyzed (Participants) | 50 | 57
Participants | 3 | 13
Statistical Analysis 1: Comparison: Fast-track Surgery vs Traditional Surgery; Test type: Superiority; p = 0.014, Chi-squared

5. Secondary Outcome: Number of Participants With Infection,
Description: infection(wound infection, lung infection, intraperitoneal infection, operation space infection)
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fast-track Surgery | Traditional Surgery
Number analyzed (Participants) | 50 | 57
Participants | 2 | 12
Statistical Analysis 1: Comparison: Fast-track Surgery vs Traditional Surgery; Test type: Superiority; p = 0.034, Chi-squared

6. Secondary Outcome: Number of Participants With Postoperative Nausea and Vomiting (PONV)
Description: it was recognized that nausea and vomiting are common side effects of surgical recovery
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fast-track Surgery | Traditional Surgery
Number analyzed (Participants) | 50 | 57
Participants | 0 | 0
Statistical Analysis 1: Comparison: Fast-track Surgery vs Traditional Surgery; Test type: Superiority; p = 1, Chi-squared

7. Secondary Outcome: Number of Participants With Ileus
Description: is a disruption of the normal propulsive ability of the gastrointestinal tract
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fast-track Surgery | Traditional Surgery
Number analyzed (Participants) | 50 | 57
Participants | 1 | 1
Statistical Analysis 1: Comparison: Fast-track Surgery vs Traditional Surgery; Test type: Superiority; p = 1, Chi-squared

8. Secondary Outcome: Number of Participants With Postoperative Haemorrhage
Description: Evidence of blood loss from drains or based on ultrasonography
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fast-track Surgery | Traditional Surgery
Number analyzed (Participants) | 50 | 57
Participants | 0 | 0
Statistical Analysis 1: Comparison: Fast-track Surgery vs Traditional Surgery; Test type: Superiority; p = 1, Chi-squared

9. Secondary Outcome: Number of Participants With Postoperative Thrombosis
Description: Evidence of blood thrombosis of participants after surgery
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fast-track Surgery | Traditional Surgery
Number analyzed (Participants) | 50 | 57
Participants | 0 | 0
Statistical Analysis 1: Comparison: Fast-track Surgery vs Traditional Surgery; Test type: Superiority; p = 1, Chi-squared

10. Secondary Outcome: PCT Calcitonin Postoperative
Description: value of calcitonin postoperative
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Fast-track Surgery | Traditional Surgery
Number analyzed (Participants) | 50 | 57
μg/L | 0.6275 (0.90827) | 0.7280 (0.89083)
Statistical Analysis 1: Comparison: Fast-track Surgery vs Traditional Surgery; Test type: Superiority; p = 0.601, t-test, 2 sided; Mean Difference (Final Values) = -0.10046, 95% CI 2-sided [-0.4819 to 0.2817], Standard Error of Mean 0.1915

11. Secondary Outcome: Cost of Surgical Therapy
Description: Cost of surgical therapy (RMB)
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: RMB
Arm/Group | Fast-track Surgery | Traditional Surgery
Number analyzed (Participants) | 50 | 57
RMB | 9703.22 (1739.157) | 9538.47 (1548.385)
Statistical Analysis 1: Comparison: Fast-track Surgery vs Traditional Surgery; Test type: Superiority; p = 0.605, t-test, 2 sided; Mean Difference (Final Values) = 164.746, 95% CI 2-sided [-465 to 794], Standard Error of Mean 317.79

ADVERSE EVENTS:
Time Frame: 6 months
Description: digestive tract fistula
Arm/Group | Fast-track Surgery | Traditional Surgery
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/57
Other Adverse Events (participants affected / at risk) | 0/50 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-01-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT02687412/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT02687412/Prot_SAP_001.pdf